CLINICAL TRIAL: NCT00080314
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Aripiprazole in the Treatment of Patients With Bipolar I Disorder With a Major Depressive Episode
Brief Title: Study of Aripiprazole in Patients With Bipolar I Disorder With a Major Depression Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-096
Record Dates: First submitted 2004-03-26; First posted 2004-03-30 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar 1 Disorder, depressed
MeSH Terms: conditions — Bipolar Disorder; Consciousness Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 10mg (2 5mg tablets), Once daily, 8 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, 0 mg, Once daily, 8 weeks.
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate flexible doses (5-30mg) of aripiprazole versus placebo in patients with bipolar depression.

ELIGIBILITY:
* ages 18-65
* Men and women, who have experienced a prior manic episode that required hospitalization, and now meet criteria for a major depressive episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change on a depression rating scale at endpoint

SECONDARY OUTCOMES:
Response rate and Clinical Global Impression scale at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (28):
  - Local Institution, Tuscaloosa, Alabama
  - Local Institution, Little Rock, Arkansas
  - Local Institution, San Diego, California
  - Local Institution, Sherman Oaks, California
  - Local Institution, Norwich, Connecticut
  - Local Institution, West Haven, Connecticut
  - Local Institution, Jacksonville, Florida
  - Local Institution, Maitland, Florida
  - Local Institution, Orlando, Florida
  - Local Insstitution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Lake Charles, Louisiana
  - Local Institution, Rockville, Maryland
  - Local Institution, Durham, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Beachwood, Ohio
  - Local Institution, Dayton, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Portland, Oregon
  - Local Institution, Media, Pennsylvania
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Lake Jackson, Texas
  - Local Institution, Wichita Falls, Texas
  - Local Institution, Arlington, Virginia
  - Local Institution, Bellevue, Washington